CLINICAL TRIAL: NCT03257735
Title: A Prospective and Observational Study of the Consistency of Gene Mutation Status Between Cerebrospinal Fluid, Blood and Tumor Tissue,and Correlation With Efficacy in Non-small Cell Lung Cancer Patients With Brain Metastases
Brief Title: A Study of the Gene Mutation Status in Cerebrospinal Fluid, Blood and Tumor Tissue of Non-small Cell Lung Cancer Patients With Brain Metastases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li-kun Chen, Chief Physician, Sun Yat-sen University
Other Study IDs: A2017-003
Record Dates: First submitted 2017-08-05; First posted 2017-08-22 (Actual); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Lung Cancer; Brain Metastases; Cerebrospinal Fluid; Next-generation Sequencing
MeSH Terms: conditions — Lung Neoplasms; Brain Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We plan to detect the patients' cerebrospinal fluid,blood and tumor tissue with the method of next-generation sequencing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: next-generation sequencing — 1. Patients' cerebrospinal fluid, blood and tumor tissue were collected within 3 days before treatment at diagnosis.
  2. Patients' cerebrospinal fluid and blood were extracted at the time of first evaluation of efficacy after treatment (TKI began after 1 month or chemotherapy after 2 cycles).
  3. Patients' cerebrospinal fluid and blood were extracted at first time of tumor progression，and re-biopsy of tumor tissue was done as much as possible.
  All the samples were tested by next-generation sequencing.

SUMMARY:
Primary lung cancer is one of the most common malignancies in China, with 57 percent of patients being diagnosed at advanced stage. At present, advanced lung cancer has entered the era of precise treatment. So it is very important to determine the gene mutation status of the tumor and prescribe drugs at the targets. Liquid biopsy is a suitable alternative when tumor tissues are difficult to obtain. Liquid biopsy technique refers to the use of human body fluid as a sample source to detect the information of related diseases, including blood, urine, saliva and cerebrospinal fluid. It is non-invasive, fast and simple, and can avoid the problem of insufficient sample size and support for repeated sampling to continuously monitor disease.

With the increasing incidence of lung cancer and the development of diagnosis and treatment technology, the survival period of patients has been extended, and the incidence and diagnosis rate of the brain metastasis of lung cancer have increased year by year. The brain metastasis of lung cancer is the most common type of brain metastatic tumor. The incidence rate is about 40-50%, and the prognosis is poor--the natural median survival period is about 1-2 months. Because of the impractical intracranial tumor biopsy and very low level of DNA in peripheral blood, cerebrospinal fluid, which makes close contact with brain tumors, becomes potential available samples. Several studies have shown that genetic testing of cerebrospinal fluid is feasible. Therefore, this study aims to test the cerebrospinal fluid, blood and tissue by the latest second-generation sequencing technology at different time points, to dynamically monitor the gene mutation status of cerebrospinal fluid, blood and tissue, to explore the role of cerebrospinal fluid biopsy in the diagnosis and treatment of non-small cell lung cancer with brain metastases.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged over 18 and less than 75 years old
2. The estimated survival period is greater than 12 weeks
3. ECOG score is less than 2
4. Histological diagnosis is non-small cell lung cancer, and there are enough tissue specimens for lung cancer related gene detection
5. The brain metastasis is confirmed by brain MRI, and the first line treatment of brain metastasis was considered as chemotherapy or target therapy
6. There must be at least one evaluable lesion based on the criteria of RECIST 1.1 (maximum diameter at least 10mm on spiral CT and MRI)
7. Patients are tolerable for lumbar puncture with no contraindication
8. Patients are able to comply with the research requirements and follow-up procedures
9. Patients must sign the informed consent prior to the beginning of any substantive test procedure (informed consent is subject to approval of the independent ethics committee)

Exclusion Criteria:

1. Brain metastases were treated
2. Intracranial symptoms were obvious, and radiotherapy/surgery was considered in the first line treatment
3. Histological specimens are not enough to detect lung cancer related genes
4. Patients were suffering from other types of malignancy
5. Patients have any contraindications of lumbar puncture
6. Patients have any uncontrolled systemic disease, including active infection, uncontrolled high blood pressure, diabetes, unstable angina and congestive heart failure, myocardial infarction (1 year) before the start of treatment, severe arrhythmia that needs drugs therapy, coagulant function abnormality, liver or kidney or metabolic disease
7. Pregnant and lactating pregnant women
8. Patients were not willing to be followed up

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were histologically confirmed with NSCLC and identified with new brain metastases by MRI.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-05-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline gene mutation status at 2 months | 2 months
  compare the gene mutation status of cerebrospinal fluid,blood and tumor tissue at baseline and after the first session
Change from second line gene mutation status at 6 months | 6 months
  compare the gene mutation status of cerebrospinal fluid,blood and tumor tissue after the first session and at the time of tumor progression

SECONDARY OUTCOMES:
PFS | From date of randomization until the date of first documented progression or date of death from any cause,whichever came first,assessed up to 60 months.
  progression-free survival
OS | From date of randomization until the date of death from any cause,assessed up to 60 months
  overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Likun Chen, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data are not available to others.

REFERENCES:
- [Derived] Li M, Chen J, Zhang B, Yu J, Wang N, Li D, Shao Y, Zhu D, Liang C, Ma Y, Ou Q, Hou X, Chen L. Dynamic monitoring of cerebrospinal fluid circulating tumor DNA to identify unique genetic profiles of brain metastatic tumors and better predict intracranial tumor responses in non-small cell lung cancer patients with brain metastases: a prospective cohort study (GASTO 1028). BMC Med. 2022 Nov 14;20(1):398. doi: 10.1186/s12916-022-02595-8. PMID 36372873